CLINICAL TRIAL: NCT03824080
Title: A Phase II Study Evaluating the Efficacy and Safety of Bemcentinib in Patients With Myelodysplastic Syndromes Failing Standard of Care Therapy
Brief Title: Evaluating the Efficacy and Safety of Bemcentinib in Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Groupe Francophone des Myelodysplasies (Other); Amsterdam UMC, location VUmc (Other); BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BERGAMO_GWT12470_2017
Record Dates: First submitted 2019-01-02; First posted 2019-01-31 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Acute Myeloid Leukemia; High-risk Myelodysplastic Syndrome; Low-risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — bemcentinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bemcentinib (Experimental): Bemcentinib will be self-administered orally (fasted) at a dose mentioned above for a total of at least 4 cycles without a treatment-free period in between.
  Responding patients (as per criteria of European LeukaemiaNet and International MDS working Group (2006)) are eligible for up to 5 additional cycles according to the maintenance daily dosing of 2 x 1 capsules of 100 mg for each 28 days cycle (up to 9 cycles in total).
  Interventions: Drug: Bemcentinib

INTERVENTIONS:
Drug: Bemcentinib — Bemcentinib will be self-administered orally (fasted) at a dose mentioned above for a total of at least 4 cycles daily.
  Responding patients (defined as at least stable disease) are eligible for up to 5 additional cycles according to the maintenance daily dosing of 2 x 1 capsules of 100 mg for each 28 days cycle (up to 9 cycles in total).

SUMMARY:
This is an open-label, single-arm multicenter, phase II study. The primary objective is to assess the efficacy of bemcentinib (BGB324) a highly selective inhibitor of the AXL receptor tyrosine kinase for the treatment of AML and MDS patients failing or being refractory to first line hypomethylating agent (HMA) treatment. Furthermore, safety, disease progression, treatment failure will be assessed. A total of 43 patients will be included in the trial.

DETAILED DESCRIPTION:
Novel treatment options in patients with MDS or AML are urgently needed; treatment has not changed significantly over the past decades and survival is still dismal, especially in elderly patients not capable for an allogeneic stem cell transplantation and failing first line treatment with hypomethylating agents. Axl, a member of the Tyro3, Axl, Mer (TAM) receptor family, mediates proliferation and survival of leukemic cells and is upregulated upon cytostatic treatment. In addition, leukemic cells induce expression of the Axl ligand growth arrest-specific gene 6 (Gas6) in bone marrow stroma cells, which further amplifies their growth and therapy resistance. selective inhibition of Axl signaling by the small molecule Axl inhibitor bemcentinib blocked leukemic proliferation in vitro and in mouse models. It was shown that a blockade of the Gas6/Axl signaling axis by R428 (bemcentinib) significantly impaired MDS growth in an ex-vivo stroma-dependent co-culture setting using patient-derived primary material. These effects were especially observed in the CD34+ MDS stem cell compartment. A persistence of this stem cell compartment is expected to underlie drug resistance and/or drive disease progression in MDS. Thus, Axl represents a potential novel target in higher risk MDS and AML.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male and female ≥ 18 years at the first screening
* Must be able to adhere to the study visit schedule and other protocol requirements
* Initial diagnosis of AML or MDS according to WHO 2016 classification
* At least one cytopenia (ANC < 1800/μL or platelet count < 100,000/μL or hemoglobin < 10 g/dL)
* Failure to achieve complete or partial response or hematological improvement after at least six (azacitidine) or four (decitabine) 4-week treatment cycles administered during the past two years OR Relapse after initial complete or partial response or hematological improvement observed after at least six (azacitidine) or four (decitabine) 4-week treatment cycles administered during the past two years OR Intolerance to treatment with HMAs during the past two years
* Not eligible for allogeneic stem cell transplantation
* ≥ 5% bone marrow blasts at central morphology
* Off all other treatments for AML/MDS for at least four weeks; G-CSF and erythropoietin are - allowed before and during the study as clinically indicated
* ECOG performance status of 0-2
* Availability of blood counts and transfusion events for previous 2 months

Exclusion Criteria:

* Prior intensive chemotherapy for MDS or AML
* Radiotherapy or chemotherapy within the 14 days prior to the first dose of Bemcentinib being administered (other than hydroxyurea)
* History of the following cardiac conditions:
* Congestive cardiac failure of > Class II severity according to the NYHA (defined as symptomatic at less than ordinary levels of activity)
* Ischemic cardiac event including myocardial infarction within 3 months prior to first dose
* Uncontrolled cardiac disease, including unstable angina, uncontrolled hypertension (i.e. sustained systolic BP >140 mmHg or diastolic BP >90 mmHg), or need to change medication within 6 weeks of provision of consent due to lack of disease control
* History or presence of sustained bradycardia (≤ 60 BPM), left bundle branch block, cardiac pacemaker or ventricular arrhythmia. (Note: Patients with a supraventricular arrhythmia requiring medical treatment, but with a normal ventricular rate are eligible )
* Family history of long QTc syndrome; personal history of long QTc syndrome or previous drug-induced QTc prolongation of at least Grade 3 (QTc > 450 ms at baseline)
* Abnormal left ventricular ejection fraction on echocardiography or Multi Gated Acquisition Scan (MUGA) (less than the lower limit of normal for a patient of that age at the treating institution or < 45 %, whichever is lower)
* Current treatment with any agent known to cause Torsades de Pointes which cannot be discontinued at least five half-lives or two weeks prior to the first dose of study treatment. Please see Appendix XI for list of relevant medications
* Screening 12-lead ECG with a measurable QTc interval according to Fridericia's correction > 450 ms
* Ongoing infection requiring systemic treatment. Patients who are on prophylactic antimicrobials or who have been afebrile for 48 hours following the initiation of antimicrobials are eligible
* Inadequate liver function as demonstrated by serum bilirubin ≥ 1.5 times the upper limits of normal range (ULN) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 times the ULN (or ≥ 5 times the ULN for AST or ALT in the presence of liver involvement by leukemia)
* Inability to tolerate oral medication
* Existing gastrointestinal disease affecting drug absorption such as celiac disease or Crohn's disease
* Known lactose intolerance, congenital lactase deficiency, galactosemia, Glucose-galactose malabsorption
* Treatment with any of the following: histamine receptor 2 inhibitors, proton pump inhibitors or - antacids within 3 days or 5 half-lives of administration of BGB234, whichever is longer
* Treatment with more than 40 mg prednisolone (or equivalent dose of systemic corticosteroid) which cannot be discontinued up to one week prior to starting Bemcentinib
* Treatment with medications which are predominantly metabolized by CYP3A4 and have a narrow therapeutic index (examples of medication are in the appendix X15.10.2)
* Previous bowel resection that would interfere with drug absorption
* Impaired renal function as demonstrated by a creatinine clearance of < 30 mL/min determined by Cockcroft-Gault formula
* Unresolved CTCAE > Grade 2 toxicity (other than stable toxicity) from previous anticancer therapy excluding alopecia
* Any evidence of severe or uncontrolled systemic conditions (e.g., severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
* Known active, uncontrolled central nervous system (CNS) disease including CNS leukemia
* Known active infection with human immunodeficiency virus (HIV), hepatitis B or C viruses - screening for viral infections is not required for entry to this study
* Major surgery within 28 days prior to the start of Bemcentinib - excluding skin biopsies and procedures for insertion of central venous access devices
* Patients who are unwilling to follow strict highly effective contraception requirements including combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion2, vasectomised partner, sexual abstinence, surgical sterilization)) before entry and throughout the study. Female patients with reproductive potential who do not have a negative urine ß-HCG pregnancy test at screening and not more than 3 days prior to initiation of treatment
* Female patients who are lactating
* Exclusion periods from other studies or simultaneous participation in other clinical studies (excluding non-interventioneal studies/registries)
* Criteria which in the opinion of the investigator precluded participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety
* Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g. employee or student of the investigational site)
* Subject is an employee of GWT-TUD GmbH or participating study groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy of Bemcentinib for the treatment of AML and MDS patients failing or being refractory to hypomethylating agent treatment | 17 weeks
  Overall hematological response rate

SECONDARY OUTCOMES:
Disease progression | up to 9 month
  Disease progression measured by increase of bone marrow blasts
Treatment failure | up to 9 month
  Time to treatment failure
Toxicity measured by NCI CTCAE 5.0 | up to 9 month
  toxicity measured by NCI CTCAE 5.0

OTHER OUTCOMES:
Immunophenotyping | up to 9 month
  Evaluating the role of potential biomarkers via flow-bases immunophenotyping of MDS and AML samples
Biomarker analysis of Axl/Gas6 | up to 9 month
  pAxl Analysis, gene expression and Axl immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof., Principal Investigator — Universitätsklinikum Leipzig
Locations (8):
- France (3):
  - CHU Hôtel Dieu Service d'Hématologie Clinique, Nantes, Nantes Cedex 1
  - Service d'Hématologie Séniors, Paris, Paris 7
  - Hôpital Archet 1 Service d'Hématologie Clinique, Nice
- Germany (4):
  - Universitätsklinikum Dresden, Dresden
  - Marien Hospital GmbH, Düsseldorf
  - Universitätsklinikum Leipzig, Leipzig
  - Technische Universität München, Klinikum rechts der Isar, Munich
- VU University Medical Center, Amsterdam, Netherlands